CLINICAL TRIAL: NCT01111318
Title: Pharmacokinetics, Safety and Tolerability of BI 10773 50 mg Single Dose in Male and Female Subjects With Different Degrees of Liver Impairment (Child-Pugh Classification A, B and C) as Compared to Male and Female Healthy Subjects (a Non-blinded, Parallel Group Study of Phase I)
Brief Title: Pharmacokinetics of Empagliflozin (BI 10773) in Patients With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.13; 2009-017202-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Hepatic Insufficiency; Healthy
MeSH Terms: conditions — Hepatic Insufficiency | interventions — empagliflozin

ARMS (1):
- BI 10773 (Experimental): 50 mg single dose
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — 2 tablets BI 10773 25 mg single dose

SUMMARY:
The main objective of this study is to assess the effect of mild, moderate and severe hepatic impairment on the pharmacokinetics, safety and tolerability of BI 10773 following oral administration of BI 10773 as a single dose.

ELIGIBILITY:
Inclusion criteria:

Healthy males and females. Hepatically impaired male and female subjects. Age: 18 - 75 years, BMI: 18-34 kg/m2 Creatinine clearance >80 mL/min (except for patients with severe hepatic impairment, see exclusion criteria.

Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

Healthy subjects (group 1)

1. Significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders as judged by the investigator.
2. Relevant gastrointestinal tract surgery.
3. Diseases of the central nervous system or psychiatric disorders or relevant neurological disorders.
4. History of relevant orthostatic hypotension, fainting spells or blackouts; systolic blood pressure < 100 or > 160 mm Hg, diastolic blood pressure < 60 or > 100 mm Hg, pulse rate < 50 or > 100 1/min.
5. Chronic or relevant acute infections.
6. History of allergy/hypersensitivity.
7. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial.
8. Use within 10 days prior to administration or during the trial of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation
9. Participation in another trial with an investigational drug within 2 months after a multiple dose study or within 1 month after a single dose study.
10. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day).
11. Inability to refrain from smoking when confined to the study site on trial days.
12. Alcohol abuse, drug abuse.
13. Veins unsuited for iv puncture on either arm.
14. Blood donation (more than 100 mL within four weeks prior to administration or during the trial).
15. Excessive physical activities (within 48 hours prior to trial or during the trial).
16. Any laboratory value outside the reference range that is of clinical relevance.
17. Inability to comply with dietary regimen of study centre.
18. Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

    Hepatically impaired subjects (group 2-4):
19. Decompensated gastrointestinal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
20. For patients with severe liver impairment (Child-Pugh C): Severe concurrent renal dysfunction (e.g., due to hepato-renal syndrome) and a creatinine clearance <40mL/min.
21. Relevant gastrointestinal tract surgery.
22. Diseases of the central nervous system or psychiatric disorders or relevant neurological disorders.
23. Chronic or relevant acute infections.
24. History of allergy/hypersensitivity.
25. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial.
26. Use within 10 days prior to administration or during the trial of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation. Co-medication known to inhibit or induce P-glycoprotein (such as quinidine, cyclosporine, amiodarone) is not allowed. In dubious cases, a case by case decision will be made after consultation with the sponsor.
27. Participation in another trial with an investigational drug within 2 months after a multiple dose study or within 1 month after a single dose study.
28. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day).
29. Inability to refrain from smoking when confined to the study site on trial days.
30. Alcohol abuse, Drug abuse.
31. Blood donation (more than 100 mL within four weeks prior to administration or during the trial).
32. Excessive physical activities (within 48 hours prior to trial or during the trial).
33. Clinically relevant laboratory abnormalities.
34. Inability to comply with dietary regimen of study centre.
35. Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

    For female subjects of all groups:
36. Pregnancy
37. Positive pregnancy test
38. No adequate contraception during the study and until 2 months after study completion.
39. Lactation period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.13.40001 Boehringer Ingelheim Investigational Site, Timișoara, Romania

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy: Single oral dose of empagliflozin (empa) 50mg (2 tablets of 25mg) following an overnight fast, for healthy subjects with normal liver function who matched the hepatically impaired subjects with regard to age and weight.
- Mild: Single oral dose of empagliflozin (empa) 50mg (2 tablets of 25mg) following an overnight fast, for patients with mild liver impairment defined by Child-Pugh class A.
- Moderate: Single oral dose of empagliflozin (empa) 50mg (2 tablets of 25mg) following an overnight fast, for patients with moderate liver impairment defined by Child-Pugh class B.
- Severe: Single oral dose of empagliflozin (empa) 50mg (2 tablets of 25mg) following an overnight fast, for patients with severe liver impairment defined by Child-Pugh class C.
Period: Overall Study
Arm/Group | Healthy | Mild | Moderate | Severe
Started | 12 | 8 | 8 | 8
Completed | 12 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Mild | Moderate | Severe | Total
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (9.2) | 57.0 (6.9) | 51.0 (8.5) | 53.9 (9.6) | 53.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 3 | 4 | 19
  Male | 4 | 4 | 5 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
  The standard deviation is actually the coefficient of variation. The 'measured values' show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: Pre-dose and 20minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 72h and 96h after drug administration
Population: Pharmacokinetic (PK) set included all subjects who were documented to have taken the investigational treatment, who provided at least one observation for at least one primary PK endpoint, without important protocol violations relevant to the evaluation of PK, provided no vomiting occurred at or before two times median tmax.
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
nmol*h/L | 10800 (22.6) | 13800 (38.6) | 16100 (26.2) | 19000 (27.1)
Statistical Analysis 1: Comparison: Healthy vs Mild; Ratio calculated as mild divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 123.15, 90% CI 2-sided [98.89 to 153.36], Standard Deviation 29.0 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Healthy vs Moderate; Ratio calculated as moderate divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 146.97, 90% CI 2-sided [118.02 to 183.02], Standard Deviation 29.0 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Healthy vs Severe; Ratio calculated as severe divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 174.70, 90% CI 2-sided [140.29 to 217.55], Standard Deviation 29.0 — Standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma.
  The standard deviation is actually the coefficient of variation. The 'measured values' show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
nmol/L | 1370 (33.9) | 1430 (36.8) | 1660 (26.4) | 1970 (22.1)
Statistical Analysis 1: Comparison: Healthy vs Mild; Ratio calculated as mild divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 103.81, 90% CI 2-sided [82.29 to 130.95], Standard Deviation 30.7 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Healthy vs Moderate; Ratio calculated as moderate divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 123.31, 90% CI 2-sided [97.74 to 155.55], Standard Deviation 30.7 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Healthy vs Severe; Ratio calculated as severe divided by healthy; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to hepatic impairment status); Geometric mean ratio = 148.41, 90% CI 2-sided [117.65 to 187.23], Standard Deviation 30.7 — Standard deviation is actually the geometric coefficient of variation

3. Secondary Outcome: Area Under the Curve 0 to Time of Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to the time of the last quantifiable data point.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
nmol*h/L | 10700 (22.6) | 13700 (38.4) | 15800 (25.7) | 18600 (23.9)

4. Secondary Outcome: Time From Dosing to Maximum Concentration (Tmax)
Description: Time from dosing to maximum concentration of empagliflozin (empa) in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
h | 2.00 (50.1) [1.00 to 4.00] | 1.50 (73.2) [0.67 to 4.00] | 2.00 (64.4) [0.67 to 2.50] | 1.50 (48.2) [0.67 to 2.50]

5. Secondary Outcome: Terminal Rate Constant (λz)
Description: Terminal rate constant in plasma.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
1/h | 0.0414 (41.6) | 0.0404 (23.5) | 0.0454 (28.9) | 0.0506 (41.1)

6. Secondary Outcome: Terminal Half-Life (t1/2)
Description: Terminal half-life of empagliflozin (empa) in plasma.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
h | 19.9 (43.1) | 18.1 (25.9) | 17.1 (45.9) | 17.7 (67.4)

7. Secondary Outcome: Mean Residence Time (MRTpo)
Description: Mean residence time of empagliflozin (empa) in the body.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
h | 13.2 (31.3) | 14.4 (22.9) | 15.5 (37.2) | 15.7 (43.0)

8. Secondary Outcome: Apparent Clearance After Extravascular Administration (CL/F)
Description: Apparent clearance of empagliflozin (empa) in the plasma after extravascular administration.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
mL/min | 179 (23.9) | 150 (34.4) | 124 (30.7) | 103 (23.0)

9. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: Apparent volume of distribution during the terminal phase (λz).
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
L | 298 (39.5) | 237 (45.5) | 173 (35.0) | 144 (46.7)

10. Secondary Outcome: Amount of Empagliflozin That is Eliminated in Urine (Ae0-96)
Description: Amount of empagliflozin (empa) that is eliminated in urine over the time interval 0 to 96 hours.
  The standard deviation is actually the coefficient of variation.
Time Frame: Pre-dose and time intervals 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h and 72-96h after drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
nmol | 18400 (26.5) | 16900 (20.6) | 18500 (35.0) | 22500 (23.5)

11. Secondary Outcome: Fraction of Empagliflozin Excreted Unchanged in Urine (fe0-96))
Description: Fraction of empagliflozin (empa) excreted unchanged in urine from time points 0 to 96 hours.
  The standard deviation is actually the coefficient of variation.
Time Frame: Pre-dose and time intervals 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h and 72-96h after drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of empagliflozin
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
percentage of empagliflozin | 16.6 (26.5) | 15.2 (20.6) | 16.7 (35.0) | 20.3 (23.5)

12. Secondary Outcome: Renal Clearance After Extravascular Administration (CL R)
Description: Renal clearance of empagliflozin (empa) in plasma after extravascular administration.
  The standard deviation is actually the coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
mL/min | 28.7 (30.3) | 23.7 (48.0) | 19.9 (36.8) | 21.3 (37.1)

13. Secondary Outcome: Urinary Glucose Excretion (UGE)
Description: Urinary glucose excretion, this endpoint was measured using Ae0-96.
  The standard deviation is actually the coefficient of variation.
Time Frame: Pre-dose and time intervals 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h and 72-96h after drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 7 | 8 | 8
mg | 86600 (34.8) | 81000 (26.7) | 79700 (67.9) | 79800 (45.6)

14. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Clinical Laboratory Tests and Assessment of Tolerability by the Investigator
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, clinical laboratory tests and assessment of tolerability by the investigator. New abnormal findings or worsening of baseline conditions were reported as Adverse Events (AE).
Time Frame: Drug administration until 4 days after drug administration or end-of-study visit, up to 19 days
Population: Treated Set (TS) included all subjects who had been dispensed study medication and were documented to have taken the investigational treatment.
Measure: Number; unit: participants
Arm/Group | Healthy | Mild | Moderate | Severe
Number analyzed (Participants) | 12 | 8 | 8 | 8
participants
  Investigations: Electrocardiogram abnormal | 2 | 0 | 0 | 0
  Investigations: Nitrite urine present | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Drug administration until 4 days after drug administration or end-of-study visit, up to 19 days
Arm/Group | Healthy | Mild | Moderate | Severe
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/12 | 0/8 | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy (N=12) | Mild (N=8) | Moderate (N=8) | Severe (N=8)
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 2 | 0 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.